CLINICAL TRIAL: NCT00002155
Title: A Six-Month Safety and Antiviral Study in HIV-1 Seropositive, AZT-Experienced Patients With CD4 Counts Less Than or Equal to 50 Cells/mm3 to Evaluate MK-639 Alone Versus Zidovudine (AZT) and 3TC Versus the Combination of MK-639 With AZT/3TC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 246E; 039
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-06

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antiviral Agents; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Indinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To compare effects on CD4 counts and serum viral RNA among HIV-seropositive, zidovudine (AZT)-experienced patients in three treatment arms: indinavir sulfate ( MK-639; Crixivan ) plus AZT plus lamivudine ( 3TC ) versus MK-639 alone versus AZT/3TC.

DETAILED DESCRIPTION:
AZT-experienced patients are randomized to receive MK-639/AZT/3TC or MK-639 alone or AZT/3TC. Additionally, patients who have received < 6 months of AZT or who are intolerant but received prior 3TC or who require concomitant rifampin therapy may receive open-label MK-639.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed for all patients:

* Standard prophylaxis for opportunistic infections.
* Continuation of treatment for opportunistic infection.

Allowed for open-label study patients:

* Rifampin.

Patients must have:

* HIV positivity.
* CD4 count <= 50 cells/mm3.
* More than 6 months of prior AZT (blinded study only).

NOTE:

* Patients on the open-label study must have AZT intolerance or have < 6 months of prior AZT.

Prior Medication:

Required for blinded study patients:

* > 6 months of prior AZT.

Required for open-label study patients:

* < 6 months of prior AZT.

Allowed for open-label study patients:

* Prior 3TC.

Exclusion Criteria

Concurrent Medication:

Excluded in all patients:

* Immunosuppressants.

Excluded in blinded study patients:

* AZT, ddI, ddC, or d4T.
* Rifampin.

Excluded in open-label study patients:

* 3TC.

Prior Medication:

Excluded in all patients:

* Prior protease inhibitors.
* Investigational agents and immunomodulators within 30 days prior to study entry.
* Immunosuppressants within 2 weeks prior to study entry.

Excluded in blinded study patients:

* Any prior 3TC.
* AZT, ddI, ddC, or d4T within 2 weeks prior to study entry.

Excluded in open-label study patients:

3TC within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600

CONTACTS AND LOCATIONS:
Locations (1):
- Merck & Co Inc, Whitehouse Station, New Jersey, United States

REFERENCES:
- [Background] Gulick RM, Mellors JW, Havlir D, Eron JJ, Gonzalez C, McMahon D, Richman DD, Valentine FT, Jonas L, Meibohm A, Emini EA, Chodakewitz JA. Treatment with indinavir, zidovudine, and lamivudine in adults with human immunodeficiency virus infection and prior antiretroviral therapy. N Engl J Med. 1997 Sep 11;337(11):734-9. doi: 10.1056/NEJM199709113371102. PMID 9287228
- [Background] Hirsch M, Steigbigel R, Staszewski S, Mellors J, Scerpella E, Hirschel B, Lange J, Squires K, Rawlins S, Meibohm A, Leavitt R. A randomized, controlled trial of indinavir, zidovudine, and lamivudine in adults with advanced human immunodeficiency virus type 1 infection and prior antiretroviral therapy. J Infect Dis. 1999 Sep;180(3):659-65. doi: 10.1086/314948. PMID 10438352